CLINICAL TRIAL: NCT04320862
Title: Pandemic Response Network: Duke Community Health Watch
Brief Title: COVID-19 Pandemic Response Network
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105189
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: COVID-19; SARS-CoV-2; Coronavirus; Influenza -Like Illness; Lower Resp Tract Infection; Upper Resp Tract Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duke Health region and beyond: Individuals in the Duke Health region as well as individuals beyond the Duke Health region who have flu-like symptoms, a viral test order for COVID-19, confirmed COVID-19, or concern for exposure to COVID-19.

SUMMARY:
Coronavirus Disease 19 (COVID-19) represents an unprecedented challenge to the operations and population health management efforts of health care systems around the world. The "Pandemic Research Network (PRN): Duke Community Health Watch" study leverages technology, clinical research, epidemiology, telemedicine, and population health management capabilities to understand how to safely COVID-19. The target population is individuals in the Duke Health region as well as individuals beyond the Duke Health region who have flu-like symptoms, a viral test order for COVID-19, confirmed COVID-19, or concern for exposure to COVID-19. A subgroup of particular interest within the target population is health care workers (HCW) and families of HCW. Community members will enroll in the study electronically and for 28 days will be reminded via email or SMS to submit signs and symptoms related to COVID-19. Participants who report symptoms will be provided information about COVID-19 testing (if needed) and established mechanisms to seek care within Duke Health. Instructions for telemedicine and in-person visits, which is available publicly at https://www.dukehealth.org/covid-19-update, will be presented to participants. Participants who are unable to report symptoms independently may be contacted via telephone by Population Health Management Office (PHMO) or Clinical Events Classification (CEC) team members. Data collected through the "Pandemic Response Network (PRN): Duke Community Health Watch" study will be used for three objectives.

* First, to characterize the epidemiological features of COVID-19. Specifically, we will have a high-risk subgroup of HCW and families of HCW that we enroll.
* Second, to develop models that predict deterioration and the need for inpatient care, intensive care, and mechanical ventilation.
* Third, to develop forecast models to estimate the volume of inpatient and outpatient resources needed to manage a COVID-19 population.

The primary risk to study participants is loss of protected health information. To address this concern, all data will be stored in Duke's REDCap instance and the Duke Protected Analytics Compute Environment (PACE).

ELIGIBILITY:
Inclusion Criteria:

* flu-like symptoms
* a viral test order for COVID-19
* confirmed COVID-19
* concern for exposure to COVID-19

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals in the Duke Health region as well as individuals beyond the Duke Health region
Sampling Method: Non-Probability Sample
Enrollment: 9207 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience inpatient admission | 2 months

SECONDARY OUTCOMES:
Number of participants admitted to the intensive care unit | 2 months
Number of participants requiring mechanical ventilation | 2 months
Number of deceased participants | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Becky Smith, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No